CLINICAL TRIAL: NCT05260164
Title: Effect of BTL-899 Device for Non-invasive Lipolysis on Human Flanks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-899_CTBG200
Record Dates: First submitted 2022-02-18; First posted 2022-03-02 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Fat Burn

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HIFEM+RF (Experimental): The subjects will be enrolled and assigned into one study arm and will be required to complete four (4) treatment visits.
  Both flanks will be treated simultaneously with the BTL-899 device for 30 minutes per session.
  Interventions: Device: HIFEM+RF

INTERVENTIONS:
Device: HIFEM+RF — Combination of High-Intensity Focused Electromagnetic Field (HIFEM) and a high radio frequency (RF) field.

SUMMARY:
This study will evaluate the clinical safety and the performance of the BTL-899 device (with its 899-AP-C-4 and 899-AP-C-5 applicators) during treatment of the flanks (also known as "love handles"). The study has a single-arm, open-label, interventional design. The subjects will be enrolled and assigned into one study arm and will be required to complete four (4) treatment visits.

Both flanks will be treated simultaneously for 30 minutes per session. The flanks' fat thickness reduction will be documented by ultrasound.

At the baseline visits health status will be assessed and, if needed, additional tests will be performed. Inclusion and exclusion criteria will be verified and informed consent will be signed.

The treatment administration phase consists of four (4) treatment visits, delivered 5 - 10 days apart.

At every treatment visit after the first, prior to the procedure, the participants will be assessed for adverse effects resulting from the previous treatment(s) with the BTL-899 device.

Safety measures will include documentation of adverse events (AE) during and after the procedures.

Follow-ups visits at 1 month and 3 months after the final treatment will be held.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index (BMI) of 20 to 35 kg/m2.
* Visible excess of adipose tissue confirmed with pinch test at the flanks ("love handles") area.
* Subjects willing and able to abstain from partaking in any treatments other than the study procedure to promote body contouring and/or weight loss during study participation.
* Successful initial determination of the flanks' fat thickness by means of ultrasound.
* No procedure for fat reduction at the treated area in the last six months.
* Subjects willing and able to maintain his/her regular (pre-procedure) diet and exercise regimen without effecting a significant change of weight in either direction during study participation.
* Age between 18 and 70 years.

Exclusion Criteria:

* Electronic implants (such as intrauterine device, cardiac pacemakers, defibrillators, and neurostimulators)
* Metal implants
* Drug pumps
* Malignant tumor
* Pulmonary insufficiency
* Injured or otherwise impaired muscles in the treatment area
* Cardiovascular diseases
* Disturbance of temperature or pain perception
* Hemorrhagic conditions
* Septic conditions and empyema
* Acute inflammations
* Systemic or local infection such as osteomyelitis and tuberculosis
* Contagious skin disease
* Elevated body temperature
* Pregnancy, postpartum period, nursing
* Graves' disease
* Scars, open lesions, and wounds at the treatment area
* Abdominal hernia
* Gynecological disease incl. inflammation in the pelvis
* Hip and rib cage trauma or recent surgery of those
* Previous liposuction in the treatment area in the last six months
* Unstable weight within the last 6 months (change in weight ± 3%)
* Previous body contouring or cellulite treatments in the flanks area in the last six months
* Any other disease or condition at the investigator's discretion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2022-03-11 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Change of fat thickness in the flanks area evaluated by ultrasound | 5 months
  To gather clinical evidence that the BTL-899 device is able to induce non-invasive lipolysis when used on human flanks

SECONDARY OUTCOMES:
Evaluation of the Therapy's Safety Measured Via Therapy Comfort Questionnaire | 5 months
  Assessment the safety of the BTL-899 device when used for non-invasive lipolysis of the flanks via questionnaires filled in by the participants following each therapy session. On Numerical Analog Scale (0-10), where 0 represents 'no pain' and 10 represents 'worst possible pain' select the level of pain experienced during the treatment. The outcome will further be measured through the occurrence of adverse events or lack thereof.
Evaluation of the participants' satisfaction with the therapy evaluated via standard questionnaires | 5 months
  Majority of the treated subjects to report satisfaction (level satisfied and higher) with the therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Practice for Specialized Medical Care - Individual practice for specialized medical dermatology care Mariya Genova MD, Plovdiv, Bulgaria

IPD SHARING:
Plan to Share IPD: No